CLINICAL TRIAL: NCT02488720
Title: Longitudinal Evaluation of Amyloid Risk and Neurodegeneration - the LEARN Study. A Companion Observational Study to Anti-Amyloid Treatment in Asymptomatic Alzheimer's Disease (A4) Trial
Brief Title: Longitudinal Evaluation of Amyloid Risk and Neurodegeneration - the LEARN Study
Acronym: LEARN
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Paul Aisen, Professor, University of Southern California
Other Study IDs: ADC-051; U19AG010483 (NIH); 15-338729 (Other: Alzheimer's Association)
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cognition Disorders
Keywords: amyloid imaging; biomarkers; cognition; longitudinal; cognitive decline; observational
MeSH Terms: conditions — Cognition Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, CSF
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clinically normal older inviduals: 500 clinically normal older individuals with florbetapir positron emission tomography (PET) scan that does not show evidence of brain amyloid pathology at screening.

SUMMARY:
The LEARN study a multicenter, observational study will that will evaluate the rate of cognitive change in approximately 500 clinically normal older individuals who "screen-fail" for the A4 trial on the basis of their screening PET imaging not demonstrating evidence of elevated amyloid accumulation (Aβ negative) but meet all other A4 study eligibility criteria. This study will leverage the A4 infrastructure and maximize the data acquired in screening a large number of well-characterized older adults for the A4 trial.

The LEARN observational cohort will provide a critical comparison group for the A4 placebo arm, and future trials in preclinical AD. Although accumulating longitudinal data suggest that older individuals with elevated Aβ burden are at increased risk of cognitive decline, it is important to demonstrate a differential rate of clinical decline between Aβe ("Aβ elevated") and Aβne ("Aβ not elevated") individuals on a standardized set of clinical outcomes. Over 2000 well-characterized, highly motivated older volunteers will "screen fail" for the A4 trial. The LEARN study will follow 500 of these individuals, matched as closely as possible to the two treatment arms, in this observation cohort. The LEARN study may selectively recruit from a specific range of SUVr that fall below the threshold for "elevated amyloid" in order to support analyses of the relationship of baseline SUVr to subsequent cognitive change and amyloid accumulation. The observational cohort will be followed for 384 weeks with identical clinical/cognitive testing performed every 24 weeks, running parallel to the A4 treatment study and open label extension.

ELIGIBILITY:
Inclusion Criteria:

1. Consented to participate in the A4 study and previously met A4 demographic, cognitive and clinical criteria (e.g., Mini-Mental State Examination (MMSE); Clinical Dementia Ratin (CDR); Logical Memory test, part IIa (LMIIa); medications; medical history).
2. Has a florbetapir PET scan that falls below the Aβ threshold levels required for randomization into the treatment arms of the A4 trial.
3. In general, permitted medications should be stable for 8 weeks prior to LEARN Visit 1. Changes to medications that, in the opinion of the investigator, are not likely to impact LEARN Visit 1 assessments are permissible.
4. Has a study partner that is willing to participate as a source of information and has at least weekly contact with the subject (contact can be in-person, via telephone or electronic communication). The study partner must have sufficient contact such that the investigator feels the study partner can provide meaningful information about the subject's daily function.
5. In the investigator's opinion, is both willing and able to participate in all required procedures for the duration of the study (at least 240 weeks), including adequate literacy in English or Spanish and adequate vision and hearing to complete the required psychometric tests.

Exclusion Criteria:

1. Is receiving a prescription acetylcholinesterase inhibitor (AChEI) and/or memantine at LEARN Visit 1
2. Has current serious or unstable illness including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic, psychiatric, immunologic, or hematologic disease or other conditions that, in the investigator's opinion, could interfere with the analyses of safety and efficacy in this study.
3. Has any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or a cardiac pacemaker that is not compatible with MRI.
4. Has a LEARN Visit 1 MRI scan with results showing >4 hemosiderin deposits (definite microhemorrhages or areas of superficial siderosis); or any amyloid-related imaging abnormalities - edema/effusions (ARIA-E).
5. Has received any exclusionary medication, including those with significant central nervous system (CNS) anticholinergic effects, within 3 months prior to LEARN Visit 1 or initiated at any point after screen. A full list of exclusionary medication will be provided in the relevant procedures manual.
6. Is currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Participation in observational studies may be permitted upon review of the observational study protocol and approval by the Project Director or one of the ADCS Medical Monitors.

   For subjects participating in the optional Lumbar Puncture (LP, all of the above, plus:
7. Current use of anticoagulants, such as warfarin or dabigatran.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 500 subjects without evidence of elevated ABeta on screening PET scan. Subjects will have consented to participate in the A4 trial and previously met demographic, cognitive and clinical criteria and have an A4 screening PET scan results that fallows below the ABeta threshold levels required for randomization into the treatment arms for the A4 trials.
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of the ADCS Preclinical Alzheimer Cognitive Composite (ADCS-PACC) to Week 240 | 4.5 years

SECONDARY OUTCOMES:
Change from Baseline in Cognitive Function Index (CFI) to Week 240 | 4.5 years
Change from Baseline in Mean Composite Summary Uptake Value Ratio (SUVr) to Week 240 | 4.5 years
Change from Baseline in Cerebral Spinal Fluid (CSF) Tau Biomarkers to Week 240 | 4.5 years
Change from Baseline of Cerebrospinal Fluid (CSF) Concentrations of Amyloid Beta (Abeta) to Week 240 | 4.5 years
Change from Baseline of Volumetric Magnetic Resonance Imaging (vMRI) to Week 240 | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Reisa Sperling, MD, Study Director — Center for Alzheimer Research and Treatment Brigham and Women's Hospital
Locations (40):
- United States (40):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - VA Palo Alto HSC / Stanford School of Medicine, Palo Alto, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Wien Center for Clinical Research, Miami Beach, Florida
  - Synexus Clinical Research, Orlando, Florida
  - University of South Florida - Health Byrd Alzheimer Institute, Tampa, Florida
  - Synexus Clinical Research - The Villages, The Villages, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Beachwood, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Butler Hospital Memory and Aging Program, Providence, Rhode Island
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Result] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Result] Vos SJ, Xiong C, Visser PJ, Jasielec MS, Hassenstab J, Grant EA, Cairns NJ, Morris JC, Holtzman DM, Fagan AM. Preclinical Alzheimer's disease and its outcome: a longitudinal cohort study. Lancet Neurol. 2013 Oct;12(10):957-65. doi: 10.1016/S1474-4422(13)70194-7. Epub 2013 Sep 4. PMID 24012374
- [Result] Jack CR Jr, Knopman DS, Jagust WJ, Shaw LM, Aisen PS, Weiner MW, Petersen RC, Trojanowski JQ. Hypothetical model of dynamic biomarkers of the Alzheimer's pathological cascade. Lancet Neurol. 2010 Jan;9(1):119-28. doi: 10.1016/S1474-4422(09)70299-6. PMID 20083042
- [Result] Mormino EC, Betensky RA, Hedden T, Schultz AP, Amariglio RE, Rentz DM, Johnson KA, Sperling RA. Synergistic effect of beta-amyloid and neurodegeneration on cognitive decline in clinically normal individuals. JAMA Neurol. 2014 Nov;71(11):1379-85. doi: 10.1001/jamaneurol.2014.2031. PMID 25222039
- [Result] Knopman DS, Jack CR Jr, Wiste HJ, Weigand SD, Vemuri P, Lowe V, Kantarci K, Gunter JL, Senjem ML, Ivnik RJ, Roberts RO, Boeve BF, Petersen RC. Short-term clinical outcomes for stages of NIA-AA preclinical Alzheimer disease. Neurology. 2012 May 15;78(20):1576-82. doi: 10.1212/WNL.0b013e3182563bbe. Epub 2012 May 2. PMID 22551733
- [Result] Lim YY, Pietrzak RH, Ellis KA, Jaeger J, Harrington K, Ashwood T, Szoeke C, Martins RN, Bush AI, Masters CL, Rowe CC, Villemagne VL, Ames D, Darby D, Maruff P. Rapid decline in episodic memory in healthy older adults with high amyloid-beta. J Alzheimers Dis. 2013;33(3):675-9. doi: 10.3233/JAD-2012-121516. PMID 23001710
- [Derived] Dubbelman MA, Liu A, Donohue MC, Langford O, Raman R, Rentz DM, Amariglio R, Sperling RA, Aisen PS, Marshall GA; as the A4 Study team. Changes in Daily Functioning in Association With Tau and Amyloid Among Unimpaired Older Adults With and Without Elevated Amyloid. Neurology. 2025 Jun 24;104(12):e213775. doi: 10.1212/WNL.0000000000213775. Epub 2025 May 29. PMID 40440591
- See also: Alzheimer's Therapeutic Research Institute — https://keck.usc.edu/atri/research/studies/